CLINICAL TRIAL: NCT05085483
Title: Efficacy of an Orally Administrated Nutritional Ketogenic Supplement, for the Prevention of Episodic Migraine: a Randomized, Double-blind, Placebo-controlled, Cross-over Trial
Brief Title: Ketone for Migraine Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Healint Pte Ltd (Unknown); Diex Research Sherbrooke Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20.08.NRC
Record Dates: First submitted 2021-10-18; First posted 2021-10-20 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (one month) (Experimental): Nutritional Ketogenic Supplement (NKS) 2 x 12 g of EKS/day
  Interventions: Dietary Supplement: Nutritional Ketogenic Supplement
- Placebo (one month) (Placebo Comparator): Isocaloric placebo supplement
  Interventions: Dietary Supplement: Isocaloric placebo supplement

INTERVENTIONS:
Dietary Supplement: Nutritional Ketogenic Supplement — This trial has 5 steps: (1) a 4-week run-in baseline; (2) a 4-week intervention phase to either active or placebo (3) a 4-week phase of washout; (4) the cross-over to the second 4-week active or placebo phase; (5) a 4-week follow-up.
  Arms: Active intervention (one month)
Dietary Supplement: Isocaloric placebo supplement — Isocaloric placebo supplement
  Arms: Placebo (one month)

SUMMARY:
Efficacy of a nutritional ketogenic supplement (NKS) in reducing the number, intensity, and duration of migraine headaches in episodic migraine patients.

DETAILED DESCRIPTION:
The KEMIP study is a randomized, placebo-controlled, double-blind, full cross-over, study to test the efficacy of NKS at reducing migraine days per month (MDM) compared to placebo in episodic migraine participants.

Participants will prompted to enter data on migraine headache features (duration, pain intensity, medication use, symptoms) and product intake in an eDiary every day throughout the course of the study.

Each participant will complete five steps of 1 month each: (1) baseline evaluation; (2) NKS/placebo intake; (3) washout & cross-over; (4) NKS/placebo intake; (5) follow-up

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years who have previously been diagnosed with migraine, with or without aura, in accordance with the ICHD-3 Classification criteria;
* Have an estimated frequency of 5 to 14 MDM in each of the 3 months prior to enrolment;
* In principle, agree at the beginning (virtual call V0) to adequately complete a headache electronic diary (e-Diary) on at least 24 days out of the 28 days in the run-in baseline period;
* In practice, adequately complete by the end of V1 a headache eDiary on at least 24 days out of the 28 days in the run-in baseline period;
* Agree to refrain from initiating or changing the type, dosage, or frequency of any prophylactic medications against migraine, and any treatments for indications other than migraine that in the opinion of the clinician may interfere with the study objectives, e.g. antidepressants, anticonvulsants, beta-blockers, etc. for the duration of the study;
* Women of childbearing potential must agree to use a medically effective form of contraception, unless they can confirm they've had bilateral tubal ligation or that their male partner has had a vasectomy (provided that the partner is the sole sexual partner of the trial participant and that the vasectomised partner has received medical assessment of the surgical success). Medically effective forms of contraception include hormonal methods, such as the contraceptive pill or implant (stable use for at least 3 months prior to enrolment), an intrauterine device (IUD) in use at least 30 days before enrolment, or barrier methods such as diaphragm plus spermicide or condom plus spermicide, in use at least 14 days before enrolment. In circumstances in which hormonal methods may interfere with the action of the IP or placebo, or in which the use of spermicides may increase the risk of transmission of disease, a double-barrier method is recommended.
* Agree to refrain from making any drastic changes to their usual diet for the duration of the study, particularly periods of fasting;
* Have a smartphone with Android or mobile operating system version compatible with eDiary;
* Able to provide informed consent

Exclusion Criteria:

Under ketogenic diet, or using exogenous ketone supplements, e.g. medium chain triglycerides (MCT) 1 month prior to the initiation of the study or during the study;

* Patients using regular high dose of Vitamin B3, calcium (>1 g/day) or magnesium (>350 mg/day) supplements 1 month prior to the initiation of the study or during the study;
* Suffer from other primary (e.g. tension-type headache, trigeminal autonomic cephalalgias, other primary headache disorders) or secondary headaches (e.g. headaches attributed to trauma or injury, vascular or non-vascular intracranial disorders, substances or their withdrawal, infections, alterations of homeostasis), hemiplegic migraine;
* Pregnancy or intending to become pregnant, or is of childbearing potential and has not had tubal ligation, has a male partner who has not had a successful vasectomy, and is unwilling to use a medically effective form of contraception, i.e. oral contraceptive pills, injectable, or implantable contraceptive; intrauterine device; or double-barrier method (e.g. diaphragm and condom), or is lactating during the study duration. In addition, women of child-bearing potential on hormone-based contraception should not intend to stop or change their contraceptive for the duration of the study;
* Significant medical history, for example diabetes mellitus, renal stones, kidney and liver failure, somatic or psychiatric conditions, uncontrolled hypertension or medicated for hypertension, known hypercalcemia, history of or current cardiovascular disease, chronic gastrointestinal (GI) disease or intestinal malabsorption, or other illness, disease or syndrome which the investigators deem unsuitable to participate in the study;
* Significant medication history, for example use of corticosteroids in format of oral or injectable;
* Vaccination planned 2 weeks prior the start of the study, or during the study;
* Patients following a sodium-restricted diet;
* History of chronic alcohol or substance misuse;
* Previously diagnosed food allergy;
* Is participating in another clinical trial or has participated in a clinical trial the preceding month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in MDM versus placebo | 1 month
  Headache eDiary will be used to record the change in monthly migraine frequency according to ICHD-3 guidelines. The headache diary captures information on date, time of onset and resolution, distinction of migraine from headache based on symptoms, pain intensity and use of acute medication

SECONDARY OUTCOMES:
Mean change from baseline in the number of headache days of any severity (headache, migraine or probable migraine, and migraine attacks) | 1 month
Proportion of responders: responders are defined as patients who had a greater than 50%, 75% or 100% reduction in MDM | 1 month
Reduction in the use of acute medication for migraine | 1 month
Mean change from baseline in migraine intensity measured with a numerical rating scale from 1 to 10; | 1 month
Mean change from baseline in the average migraine duration | 1 month
Incidence, severity and relatedness of adverse events | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ginette Girard, MD, Principal Investigator — Diex Research Sherbrooke Inc.
Locations (1):
- Diex Research Sherbrooke Inc., Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No